CLINICAL TRIAL: NCT04542096
Title: Real Time Evaluation of Dynamic Changes of the Lungs During Respiratory Support of Very Low Birth Weight (<1500 g) Neonates Using Electric Impedance Tomography
Brief Title: Real Time Evaluation of Dynamic Changes of the Lungs During Respiratory Support of VLBW Neonates Using EIT
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Arunas Liubsys, Arūnas Liubšys MD, PhD, Vilnius University
Other Study IDs: EIT-1
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2022-11

CONDITIONS: RDS - Infants; RDS of Prematurity; Respiratory Failure; Prematurity; Very Low Birth Weight Infant
Keywords: electrical impedance tomography
MeSH Terms: conditions — RDS - infants; Respiratory Distress Syndrome In Premature Infants; Respiratory Insufficiency; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group1: Patients receiving invasive respiratory therapy (intubated)
  Interventions: Device: Lung electrical impedance tomography monitoring
- Group2: Patients receiving non-invasive respiratory therapy.
  Interventions: Device: Lung electrical impedance tomography monitoring

INTERVENTIONS:
Device: Lung electrical impedance tomography monitoring — A belt for recording changes in electrical impedance in the skin will be fastened for the purpose of this study with no other additional procedures

SUMMARY:
Electric Impedance Tomography (EIT) is a lung monitoring technique based on the injection of small currents and voltage measurements using electrodes on the skin surface generating cross-sectional images representing impedance change in a slice of the thorax. It is a real time, radiation free, non-invasive and portable. Neonatal respiratory distress syndrome (RDS) is a respiratory disorder resulting from immaturity of the lung structure and lack of surfactant. It is one the most common conditions in premature infants. Many of these infants require either invasive or non-invasive respiratory support. The goal of the study is to investigate the dynamic changes in pulmonary aeration during assisted breathing in very low birthweight preterm infants using pulmonary electrical impedance tomography. Currently most widely used methods to assess respiratory lung function are either invasive and/or indirect (ABG, pulse oximetry, transcutaneous pCO2 measurement), lacks temporal resolution (lung ultrasound) or emit ionizing radiation (CT). EIT provides information on regional lung aeration without the aforementioned shortcomings.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks OR birthweight <1500 g.
* Need of respiratory therapy (invasive or non-invasive)
* Parental consent.

Exclusion Criteria:

* patient does not meet all of the above listed inclusion criteria
* patients with a pacemaker
* patients with skin damage/abrasions at the EIT device belt area
* newborns with significant thoracic deformity

Ages: 22 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates meeting eligibility criteria and treated in the Neonatal Intensive Care Unit will be invited to participate in the study. All subjects will be assessed, diagnosed and treated according to institutional guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the lung aeration properties of very low birth weight neonates using different respiratory therapy methods and regimens. | 1 - 5 days.
  Lung aeration and ventilation will be assessed with EIT. Several methods will be used and compared, based on pixel information of lung aeration, and pressure-volume characteristics, regional ventilation distribution and etc.

SECONDARY OUTCOMES:
To evaluate the characteristics of lung aeration during routine nursing care in preterm very low birthweight infants receiving respiratory support. | 1 - 5 days.
  Same as primary outcome.
To compare lung aeration and regional ventilation distribution between two non-invasive respiratory therapies, constant positive pressure and high-flow nasal cannula in very low birthweight neonates. | 1 - 5 days.
  Same as primary outcome

OTHER OUTCOMES:
Predict criteria and preconditions for the successful extubation using electrical impedance tomography | 3 days
  Same as primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Arūnas Liubšys, MD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University Santaros Klinikos, Vilnius, Vilnius County, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Virsilas E, Liubsys A, Janulionis A, Valiulis A. Noninvasive Respiratory Support Effects on Sighs in Preterm Infants by Electrical Impedance Tomography. Indian J Pediatr. 2023 Jul;90(7):665-670. doi: 10.1007/s12098-022-04413-8. Epub 2022 Dec 21. PMID 36539568